CLINICAL TRIAL: NCT07277725
Title: The Effect of Acupressure on Sleep Quality Among Elderly People in Institutional Care
Brief Title: Acupressure and Sleep Quality in Elderly Care
Acronym: ASEQ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duzce University (Other)
Responsible Party: Principal Investigator, ozlemakkas, Assistant Professor, Duzce University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018/25
Record Dates: First submitted 2025-11-29; First posted 2025-12-11 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Sleep Disorders
Keywords: Acupressure; Geriatric; Nursing; Aged care services; Quality of sleep; Sleep Disorder
MeSH Terms: conditions — Sleep Wake Disorders; Sleep Initiation and Maintenance Disorders | interventions — Acupressure

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to either the intervention group (receiving acupressure) or the control group (no intervention). Randomization was performed using a computer-assisted method to ensure balanced allocation between groups. Both groups were followed concurrently in a parallel design, with assessments conducted at the same time points.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants in the intervention group received acupressure therapy. Acupressure was applied to Shenmen (HT7), Neiguan (P6), and Sanyinjiao (SP6) points. Sessions were conducted three times per week, every other day, for four weeks (12 sessions in total).
  Interventions: Behavioral: Acupressure Therapy
- Control Group (No Intervention): Participants in the control group did not receive any intervention during the study period. They were assessed at the same time points as the intervention group using the Pittsburgh Sleep Quality Index (PSQI) and the Epworth Sleepiness Scale (ESS).

INTERVENTIONS:
Behavioral: Acupressure Therapy — The intervention consisted of acupressure therapy applied to Shenmen (HT7), Neiguan (P6), and Sanyinjiao (SP6) points. Sessions were administered three times per week, every other day, for four consecutive weeks, totaling 12 sessions. Each session lasted approximately 20 minutes and was performed by a trained researcher. Participants were assessed using the Pittsburgh Sleep Quality Index (PSQI) and the Epworth Sleepiness Scale (ESS) before and after the intervention
  Other Names: Manual Acupressure Therapy; Acupressure at HT7, P6, SP6 Points
  Arms: Intervention Group

SUMMARY:
This study was carried out in a prospective randomized controlled experimental design in order to evaluate the effect of acupressure on sleep quality and day sleepiness in individuals living in an elderly care center. The study sample consisted of 75 elderly individuals, 38 in experimental and 37 in control groups, who met the inclusion criteria, living in three different care institutions in Düzce. The data were collected using the Elderly Information Form, the Pittsburgh Sleep Quality Index (PSQI), and the Epworth Sleepiness Scale (ESS). Twelve sessions of acupressure were applied to the individuals in the experimental group every other day three times a week for four weeks. Acupressure was applied to Shenmen (HT7), Neiguan (P6), and Sanyinjiao (SP6) acupressure points. The PSQI and ESS were applied on the elderly in the experimental group before and after the application, and on the elderly in the control group before the application and at the end of the 12-session acupressure application in the experimental group. The PSQI and ESS were applied in both groups again one month after the last application. It was found that subjective sleep quality and sleep duration increased, sleep latency decreased, habitual sleep efficiency was regulated, and sleep disorders and daytime dysfunction declined through the application of acupressure in the elderly receiving institutional care. It was determined that the total PSQI score decreased and the quality of sleep increased in the experimental group following the application. Moreover, the ESS score and day sleepiness decreased in the experimental group following the application. Consequently, it was concluded that acupressure could be a supplementary and supportive method to be used for sleep disorders in the elderly.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years and older
* Able to provide informed consent
* Living in the nursing home during the study period
* Willing to participate in acupressure sessions and assessments
* Adequate cognitive ability to complete questionnaires (PSQI, ESS)

Exclusion Criteria:

* Severe cognitive impairment or dementia preventing questionnaire completion
* Presence of acute psychiatric disorder or severe communication difficulties
* Current use of sedative/hypnotic medications affecting sleep quality
* Severe medical conditions (e.g., terminal illness, unstable cardiovascular disease) that contraindicate participation

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 75 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Primary Outcome Measure | Baseline (pre-intervention) and 4 weeks after intervention
  Change in sleep quality assessed by the Pittsburgh Sleep Quality Index (PSQI). The Pittsburgh Sleep Quality Index (PSQI) was developed in 1989 by Buysse and colleagues to assess sleep quality. The scale provides a quantitative measure that allows the identification of "good sleep" and "poor sleep." It evaluates sleep quality, sleep quantity, the presence of sleep disturbances, and their severity over the past month. The scale consists of 24 questions, 19 of which are self-report items. The remaining 5 items are answered by a bed partner or roommate, used solely for clinical information, and are not included in the scoring. The PSQI includes seven components evaluating different aspects of sleep: Subjective Sleep Quality, Sleep Latency, Sleep Duration, Habitual Sleep Efficiency, A PSQI score of 5 or higher reflects clinically significant impairment in sleep quality. Based on these thresholds, sleep quality is categorized as good (0-4 points) or poor (5-21 points).

SECONDARY OUTCOMES:
Secondary Outcome Measure | Baseline (pre-intervention) and 4 weeks after intervention
  Change in daytime sleepiness assessed by the Epworth Sleepiness Scale (ESS). Epworth Sleepiness Scale (ESS) The Epworth Sleepiness Scale (ESS) was developed by Johns in 1991 to assess general daytime sleepiness in adults. The scale consists of 8 self-report items. The Cronbach's alpha reliability coefficient of the ESS was reported as 0.88 in individuals with sleep disorders (Johns, 1991). The ESS evaluates an individual's general level of daytime sleepiness. It assesses the likelihood of dozing off or falling asleep in 8 different everyday situations, asking participants to rate their likelihood of falling asleep on a typical day when they are not excessively tired. Each item is scored between 0 and 3, and the total score ranges from 0 to 24. A total score between 2 and 10 indicates normal daytime sleepiness, whereas a score of 11 or higher suggests increased daytime sleepiness.

CONTACTS AND LOCATIONS:
Overall Officials: Zeliha Tülek, Professor Doctor, Study Director — Istanbul University - Cerrahpasa
Locations (2):
- Turkey (Türkiye) (2):
  - stanbul University-Cerrahpaşa ,Graduate School of Health Sciences ,Department of Internal Medicine Nursing, Istanbul
  - stanbul University-Cerrahpaşa, Istanbul

IPD SHARING:
Plan to Share IPD: Yes
Plan Description: De-identified participant-level data will be shared, including:
  Pittsburgh Sleep Quality Index (PSQI) scores at baseline and 4 weeks post-intervention
  Epworth Sleepiness Scale (ESS) scores at baseline and 4 weeks post-intervention
  Demographic variables (age, sex) relevant to analysis
Supporting Information: Study Protocol, CSR
Time Frame: De-identified individual participant data (IPD) from the published thesis are already available. Specifically, data include Pittsburgh Sleep Quality Index (PSQI) scores, Epworth Sleepiness Scale (ESS) scores, and demographic variables (age, sex). Since the thesis has been published, these datasets are accessible upon request.
Access Criteria: De-identified individual participant data (IPD) and supporting documents (study protocol, statistical analysis plan, informed consent form) will be available to qualified researchers.
URL: https://tez.yok.gov.tr/UlusalTezMerkezi/tezSorguSonucYeni.jsp

REFERENCES:
- [Background] Samadi P, Alipour Z, Lamyian M. The Effect of Acupressure at Spleen 6 Acupuncture Point on the Anxiety Level and Sedative and Analgesics Consumption of Women during Labor: A Randomized, Single-blind Clinical Trial. Iran J Nurs Midwifery Res. 2018 Mar-Apr;23(2):87-92. doi: 10.4103/ijnmr.IJNMR_199_16. PMID 29628954
- [Background] Yeh CH, Kwai-Ping Suen L, Chien LC, Margolis L, Liang Z, Glick RM, Morone NE. Day-to-Day Changes of Auricular Point Acupressure to Manage Chronic Low Back Pain: A 29-day Randomized Controlled Study. Pain Med. 2015 Oct;16(10):1857-69. doi: 10.1111/pme.12789. Epub 2015 May 19. PMID 25988270
- [Background] Yeung WF, Ho FY, Chung KF, Zhang ZJ, Yu BY, Suen LK, Chan LY, Chen HY, Ho LM, Lao LX. Self-administered acupressure for insomnia disorder: a pilot randomized controlled trial. J Sleep Res. 2018 Apr;27(2):220-231. doi: 10.1111/jsr.12597. Epub 2017 Sep 8. PMID 28884877